CLINICAL TRIAL: NCT03955926
Title: Ultrasonographic Assessment of Stomach for Comparison of Antral Cross-sectional Area in Two Different Fasting Guidelines
Brief Title: Ultrasonographic Assessment of Stomach in Two Different Fasting Guidelines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunah Cho, MD (Other)
Responsible Party: Sponsor-Investigator, Eunah Cho, MD, Clinical Assistant Professor, Kangbuk Samsung Hospital
Organization: Kangbuk Samsung Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KBSMC IRB 2019-04-025-004
Record Dates: First submitted 2019-05-17; First posted 2019-05-20 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: General Anesthesia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): kept fasted from midnight until surgery
- NO-NPO group (Experimental): drink carbohydrate beverage until 2 h before surgery
  Interventions: Dietary Supplement: preoperative oral carbohydrate loading

INTERVENTIONS:
Dietary Supplement: preoperative oral carbohydrate loading — Carbohydrate beverage (12.8% carbohydrates, 50 kcal/100 mL, 290 mOsm/kg) 800 mL is given to the NO-NPO group until 2 hours before surgery
  Arms: NO-NPO group

SUMMARY:
Oral carbohydrate loading until 2 h before surgery is well known to be effective in facilitating postoperative recovery and reducing complications, by maintaining homeostasis. However, there are still concerns in implementing this as a universal fasting guideline, because of the risk of pulmonary aspiration. Therefore, we designed this study to compare the two preoperative fasting guideline: (1) keep fasted from midnight until surgery, and (2) oral carbohydrate beverage 800 mL from midnight until 2 h before surgery.

ELIGIBILITY:
Inclusion Criteria:

* adult aged from 18 to 70
* American Society of Anesthesiologists (ASA) class I or II
* absence of pregnancy
* not on lactation at the time of surgery

Exclusion Criteria:

* delayed gastric emptying (GERD, gastrointestinal disease, diabetes)
* contraindicated to NSAID or opioid
* mental disorders
* alcoholism
* drug abuse

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with indication for laparoscopic gynecologic surgery for benign or premalignant gynecologic conditions
Enrollment: 64 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Cross-sectional area of gastric antrum | 1 hour before surgery
  Cross-sectional area of gastric antrum assessed by ultrasonography

SECONDARY OUTCOMES:
Hunger score | 1 hour before surgery
  Hunger score is scored from 0 (never) to 10 (very much).
Thirst score | 1 hour before surgery
  Thirst score is scored from 0 (never) to 10 (very much).
Preoperative anxiety | 1 hour before surgery
  Preoperative anxiety is scored from 0 (never) to 10 (very much).

CONTACTS AND LOCATIONS:
Overall Officials: Eunah Cho, M.D., Principal Investigator — KangbukSamsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho EA, Huh J, Lee SH, Ryu KH, Shim JG, Cha YB, Kim MS, Song T. Gastric Ultrasound Assessing Gastric Emptying of Preoperative Carbohydrate Drinks: A Randomized Controlled Noninferiority Study. Anesth Analg. 2021 Sep 1;133(3):690-697. doi: 10.1213/ANE.0000000000005411. PMID 33591115